CLINICAL TRIAL: NCT02579395
Title: A Couples-based Approach for Increasing Physical Activity Among Adults With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-0601
Record Dates: First submitted 2015-10-09; First posted 2015-10-19 (Estimated); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Collaborative Implementation Intentions; Individual Implementation Intentions; Information Only Control Condition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- With spouse/romantic partner (Experimental)
  Interventions: Behavioral: Collaborative implementation Intentions
- Without spouse/romantic partner (Experimental)
  Interventions: Behavioral: Individual implementation Intentions
- Control (Other): No Intervention
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Collaborative implementation Intentions — With spouse/romantic partner
  Arms: With spouse/romantic partner
Behavioral: Individual implementation Intentions — Without spouse/romantic partner
  Arms: Without spouse/romantic partner
Behavioral: Control
  Arms: Control

SUMMARY:
In a 6-week experimental design, up to 90 adult couples in which one partner has Type 2 Diabetes (T2D) will be randomly assigned to either the collaborative implementation intentions (Collaborative IIs), the Individual Implementation Intentions (Individual IIs) condition, or the control condition. As this is a pilot study, randomization for the experimental groups vs the control groups will occur at a 2:1 ratio. Thus, the experimental conditions will contain up to 36 participants and the control condition will contain up to 18 participants. Adults with T2D who are living with a romantic partner, not meeting current physical activity guidelines but able and willing to begin a new physical activity (PA) routine and their partners will be assessed at baseline, 3 weeks and 6 weeks after the experimental manipulation. Partners will report on their own investment in the patient's goal and patients will report on their own PA self-efficacy. Patient's PA will be measured through self-report, partner report and accelerometers for a week prior to each survey assessment. These specific aims are planned:

AIM 1: Determine whether collaborative IIs for patient's PA lead to a greater increase in partner investment in partners of adults with T2D than do individual IIs or control.

AIM 2: Determine whether collaborative IIs for patient's PA lead to a greater increase in patient PA self-efficacy in adults with T2D than do individual IIs or control.

AIM 3: Determine whether collaborative IIs for patient's PA lead to a greater increase in patient PA in adults with T2D than do individual IIs or control.

ELIGIBILITY:
Inclusion Criteria:

* At least 21 years of age
* Able to read and understand English
* Does not meet physical activity guidelines (< 150 minutes of moderate-vigorous exercise per week) for the last 3 months* (only required of one partner)
* Diagnosed with Type 2 Diabetes* (only required of one partner)
* Married or living with a romantic partner

Exclusion Criteria:

* Medical or physical contraindications to participate in physical activity

Ages: 21 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Self-Reported Physical Activity via IPAQ | Baseline, 3 weeks, 6 weeks
  Participants will self-report their physical activity over the past week using the International Physical Activity Questionnaire (IPAQ)
Objective Physical Activity via accelerometer | Basline, 6 weeks
  Participants will wear Actigraph Accelerometers

SECONDARY OUTCOMES:
Physical Activity Self-Efficacy via a self efficacy scale | Baseline, 3 weeks, 6 weeks
  Physical activity self-efficacy will be measured using the self-efficacy for exercise scale (SEE; Resnick & Jenkins, 2000). This 9-item, self-report scale assesses participant's confidence that they could exercise three times per week for 20 minutes under various circumstances (e.g. "you had to exercise alone"; "you felt tired"). Respondents are asked to rate items on a scale from 1, (not at all confident), to 10 (extremely confident).
Physical Activity Partner Investment Scale | Baseline, 3 weeks, 6 weeks
  The Physical Activity Partner Investment Scale assesses the degree to which the partner in a couple defines the patient engaging in regular physical activity as a shared responsibility as well as the degree to which they are taking action to address barriers to the patient engaging in physical activity . The 9 items selected were modified to be specific to engaging in regular physical activity. Participants are asked to rate their agreement each item on a scale from 1 (strongly disagree) to 7 (strongly agree). Example items include "If/when my partner decides to engage in regular physical activity , the responsibility will be his or hers alone.", "My partner and I are able to have useful discussions about how to engage in regular physical activity ." and "In the long run, my partner and I are able to work together toward helping one or both of us maintain a regular physical activity routine".

CONTACTS AND LOCATIONS:
Overall Officials: Jennalee S Wooldridge, MA, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Denver, Colorado, United States